CLINICAL TRIAL: NCT00645684
Title: Clinical Use of an Absorbable Coated Suture Material in Surgery (Safil) One Layer Running(A) vs. Two-Layer Suture Technique (B)
Brief Title: Clinical Use of an Absorbable Coated Suture Material in Surgery (Safil)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aesculap AG (Industry)
Responsible Party: Dr. Erich Odermatt, Aesculap AG&Co. KG, 78532 Tuttlingen, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BBS-WV-H-0219
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Gastrointestinal Diseases; Laparotomy; Anastomosis, Surgical; Absorbable, Coated Sutures
Keywords: Gastrointestinal Anastomosis; Multicentre; Randomized controlled single-blind study; synthetic, absorbable, braided and coated suture material; Laparotomy
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): one layer running suture technique
  Interventions: Procedure: Gastrointestinal Anastomosis
- B (Experimental): two-layer suture technique
  Interventions: Procedure: Gastrointestinal Anastomosis

INTERVENTIONS:
Procedure: Gastrointestinal Anastomosis — Gastrointestinal Anastomosis with synthetic, absorbable, coated suture material using two different suture-techniques
  Other Names: SAFIL®: is a mid-term braided and coated synthetic absorbable suture made of; pure polyglycolic acid.

SUMMARY:
The purpose is to test a coated polyglycolic acid multifilament suture in gastrointestinal surgery as part of a controlled randomized single blinded parallel group trial. The applicability and safety of the strand material used in two suture techniques (2-layer suture technique vs. 1-layer running) are to be tested on the basis of handling characteristics, the operative time consumed for the construction of the 1st anastomosis, the average time of the hospital duration for both patient groups, and the frequency of postoperative complications after discharge, 1 month and a maximum of 3-4 months. The used suture units are counted and the length of sutures determined which will be an indirect measurement of the costs of suture material for the two techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, undergoing a gastrointestinal hand made one-layer running (A) or two-layer (B) anastomotic procedure where the use of synthetic absorbable surgical suture material is indicated.
* Written consent to participate in the study

Exclusion Criteria:

* Emergency patients that cannot be properly informed about the clinical trial and cannot give their written consent
* Pregnancy or lactation period
* Patients suffering from a diffuse purulent peritonitis or generalized diseases, which can have consequences for the healing of the asnastomosis (e.g. ubalanced diabetes, progressed uremia, massive hypoproteinaemia, sever jaundice, generalized intraabdominal tumor metastases, severe tumorous cachexia, severe avitaminosis, chronic liver disease.
* Patients who are undergoing a therapeutic procedure, which can have consequences for the healing of the anastomosis (e.g. treatment with corticosteroids or cytostatics, local radiation in the operating area)
* Laparoscopial Procedures
* Patients who are not willing to cooperate and legally incapacitated people

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 1998-04; Primary Completion 2001-09 (Actual); Study Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
Frequency of postoperative Complications | discharge, 1 month and a maximum of 3-4 months

SECONDARY OUTCOMES:
handling characteristics | intraoperative
Operation time to construct the first anastomosis | intraoperative
length of hospitalization | postoperative
costs of suture material | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: György Weber, MD, PhD, Principal Investigator — Medical School of University Pecs, Hungary
Locations (3):
- Hungary (3):
  - Bugat Pal Korhaz, Sebeszeti Osztaly, Gyöngyös
  - B.-A.-Z. Megyei Korhaz, Sebeszeti Osztaly, Miskolc
  - Medical School of University Pecs, Pécs